CLINICAL TRIAL: NCT04048538
Title: Preoperative Patient Education Via Animated Videos to Improve Patient Satisfaction and Reduce Complications in Head and Neck Surgery: a Randomized Controlled Study
Brief Title: Preoperative Patient Education Via Animated Videos to Improve Patient Satisfaction and Reduce Complications in Head and Neck Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Sena Turkdogan, Principal Investigator, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Precare
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Patient Satisfaction; Surgery
Keywords: patient education; surgical education; multimedia; animation; guide
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Individuals who will receive access to the animated multimedia platform prior to their surgical procedure.
  Interventions: Other: Precare
- Control Arm (Active Comparator): Individuals who will not receive access to the animated patient platform, and instead will receive the usual standard of care.
  Interventions: Other: usual standard of care

INTERVENTIONS:
Other: Precare — an innovative patient education platform using animated videos created by using up-to-date evidence-based informaiton
  Arms: Treatment Arm
Other: usual standard of care — individuals will receive treatment as per the usual standard of care
  Arms: Control Arm

SUMMARY:
This randomized control trial will compare traditional patient education methods (pamphlets, clinical visits) to the implementation of an innovated patient education platform. The purpose of the project is to determine whether the use of this animation based patient education platform prior to undergoing surgery will lead to improved patient satisfaction and quality of life.

DETAILED DESCRIPTION:
Hypothesis/Study question:

Does the implementation of an animation based patient education platform prior to undergoing surgery lead to improved patient satisfaction and quality of life?

Study objectives:

Help address patient gaps in understanding, reduce learning barriers in order for patients to make informed decisions, improve behaviors, and better partner with their health providers to attain optimal health outcomes

Methodology / Study design:

Patients will receive access to the patient education platform during the clinical visit in which they receive their diagnosis, and will be asked if they wish to enroll in the study consisting of completing questionnaires before and after their surgical procedure. Questions will inquire on levels of anxiety, patient satisfaction, knowledge retention, and platform feedback.

ELIGIBILITY:
Inclusion Criteria:

* Individuals having any of the following surgical procedure at the Jewish General Hospital over the next 12 months: head and neck cancer resection with or without reconstruction, excision of parotid lesion, thyroidectomy, parathyroidectomy, laryngectomy, or trans-oral robotic resection.

Exclusion Criteria:

* Individuals who are undergoing a surgical procedure not included in the ones listed above, or those who are having revision surgery or have previously had surgery in the otolaryngology, head and neck surgery department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 1 month post-operative
  analyzed using patient questionnaire responses

SECONDARY OUTCOMES:
Post-operative complication rate | 1 month post-operative
  analyzed using hospital data

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turkdogan S, Roy CF, Chartier G, Payne R, Mlynarek A, Forest VI, Hier M. Effect of Perioperative Patient Education via Animated Videos in Patients Undergoing Head and Neck Surgery: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Feb 1;148(2):173-179. doi: 10.1001/jamaoto.2021.3765. PMID 34967863